CLINICAL TRIAL: NCT01353963
Title: An Open Label, Non-interventional Study Of The Safety Of Desvenlafaxine Succinate (Pristiq) In The Treatment Of Major Depressive Disorder (Mdd) And Vasomotor Symptoms (Vms) Associated With Menopause In Filipino Adult Patients: A Post Marketing Surveillance Study
Brief Title: Desvenlafaxine Succinate (Pristiq): Postmarketing Surveillance Study Among Filipino Patients
Status: Terminated | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B2061038
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder; Vasomotor Symptoms
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: desvenlafaxine succinate

INTERVENTIONS:
Drug: desvenlafaxine succinate — 50 mg tablet once daily
  Other Names: Pristiq

SUMMARY:
This is a non-interventional study to review safety data on administration of desvenlafaxine succinate among Filipino patients with MDD and VMS per usual clinical practice within the first three years post commercial distribution.

DETAILED DESCRIPTION:
post marketing surveillance none

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with major depressive disorder and vasomotor symptoms secondary to menopause prescribed with desvenlafaxine succinate

Exclusion Criteria:

Hypersensitivity to desvenlafaxine succinate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with major depressive disorder and vasomotor symptoms secondary to menopause prescribed with desvenlafaxine succinate
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Philippines (3):
  - Private Clinic, Las Piñas
  - Private Clinic, Manila
  - Private Clinic, Pasay

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061038&StudyName=Desvenlafaxine%20Succinate%20%28Pristiq%29%3A%20Postmarketing%20Surveillance%20Study%20%20Among%20Filipino%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Desvenlafaxine Succinate: Participants diagnosed with major depressive disorder (MDD) or vasomotor symptoms (VMS) associated with menopause aged 18 years and above who received desvenlafaxine succinate as per the approved local product document were observed for 8 weeks in this prospective study. For MDD, the recommended dose of desvenlafaxine succinate was 50 milligram (mg) once daily and for VMS associated with menopause, the recommended dose of desvenlafaxine succinate was 100 mg once daily. Dose was adjusted solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Desvenlafaxine Succinate
Started | 13
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study medication during the observation period.
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs), or Discontinuation Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug with regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between Week 4 and up to Week 8 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Week 4 to Week 8
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 13
Participants
  Participants w ith AEs | 5
  Participants w ith SAEs | 0
  Participants discontinued due to AEs | 2

2. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Week 4.
Time Frame: Week 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 13
millimeter of mercury (mmHg)
  Change from baseline in systolic BP at Week 4 | -0.5 (8.69)
  Change from baseline in diastolic BP at Week 4 | -0.5 (9.60)

3. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Week 8.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 11
millimeter of mercury (mmHg)
  Change from baseline in systolic BP at Week 8 | -0.7 (7.06)
  Change from baseline in diastolic BP at Week 8 | -1.8 (13.28)

4. Primary Outcome: Change From Baseline in Heart Rate at Week 4.
Time Frame: Week 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 13
beats per minute (bpm) | 1.9 (4.50)

5. Primary Outcome: Change From Baseline in Heart Rate at Week 8.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 11
bpm | 0.6 (5.59)

6. Primary Outcome: Change From Baseline in Weight at Week 4.
Time Frame: Week 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 13
kilogram (kg) | 0.1 (1.61) [-4 to 3]

7. Primary Outcome: Change From Baseline in Weight at Week 8.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Desvenlafaxine Succinate
Number analyzed (Participants) | 11
kg | 0.5 (1.69) [-2 to 3]

ADVERSE EVENTS:
Time Frame: Week 4 to Week 8
Arm/Group | Desvenlafaxine Succinate
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desvenlafaxine Succinate (N=13)
Libido decreased (Psychiatric disorders) | 1 (1)
Ejaculation delayed (Reproductive system and breast disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the low number of subjects with data available, only descriptive summaries have been presented. The outcomes measures were prioritized as per study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.